CLINICAL TRIAL: NCT06015256
Title: Characterization of Natural Killer Cells in Severe Asthma Patients in Comparison With Control Subjects: Identification of Biomarkers, Response During Virus-induced Exacerbations, and Interaction With Bronchial Epithelial Cells
Brief Title: Characterization of Natural Killer Cells in Severe Asthma Patients in Comparison With Control Subjects
Acronym: NKAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C21-75; 2022-A00651- 42 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-07-10; First posted 2023-08-29 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Asthma Acute
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Severe uncontrolled asthma in exacerbation (Other)
  Interventions: Biological: blood sample
- Severe uncontrolled asthma excluding exacerbation (Other)
  Interventions: Biological: blood sample
- Severe controlled asthma (Other)
  Interventions: Biological: blood sample
- Healthy volunteers (control group) (Other)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — Blood sample (56mL) taken in a heparin tube

SUMMARY:
Asthma is a common chronic bronchial disease affecting 300 million people worldwide. The disease can be severe when it is not managed properly or when it is not controlled by treatments. Asthma is characterized by bronchial inflammation, bronchial hyperreactivity and tissue remodeling. Symptoms include episodes of coughing, dyspnoea and wheezing in relation with bronchial obstruction. The evolution is marked by the occurrence of exacerbations (increase of symptoms), most often triggered by viral infections, mostly due to rhinoviruses. The treatment of asthma is based on inhaled corticosteroid therapy sometimes combined with other treatments that help control the majority of asthma. However, about 10% of patients suffer from persistent symptoms despite these treatments.

Natural killer (NK) cells are important actors of the antiviral innate immune response and are present in high numbers in the lungs. However, their role in severe asthma and its virus-induced exacerbations is unknown.

The purpose of this work is to characterize NK cells in severe asthma in order to identify molecules expressed differently from control subjects. The goal is to assess whether these molecules could be potential biomarkers of a severe asthma subtype, also known as the endotype, and/or be the molecular control for exacerbation. The advantage of identifying biomarkers for inflammatory diseases lies in their usefulness in establishing a correct diagnosis, monitoring the progress of the disease and the effectiveness of treatments. The secondary objectives are to characterize the activation of NK cells in response to in vitro rhinovirus infection of different types, in monoculture or in a model of interaction with a bronchial epithelium, and identify one or more molecules involved in the interaction between bronchial epithelial cells and NK cells.

ELIGIBILITY:
Inclusion Criteria:

Cases asthma controlled, uncontrolled excluding exacerbation, uncontrolled asthma exacerbation, and healthy volunteers:

* Consent form read, understood, approved and signed before any study procedure
* Membership of a social security scheme or beneficiary of such a scheme
* Patient aged over 18

Cases asthma controlled, uncontrolled excluding exacerbation, uncontrolled exacerbation:

- Diagnosis of severe asthma confirmed by a respirologist at an expert centre

Case asthma controlled:

- Asthma control confirmed by a lung specialist from an expert centre

Case uncontrolled asthma excluding exacerbation:

- Uncontrolled asthma confirmed by a lung specialist from an expert centre

Case uncontrolled asthma with exacerbation:

- Current exacerbation

Exclusion Criteria:

Cases asthma controlled, uncontrolled excluding exacerbation, uncontrolled asthma exacerbation, and healthy volunteers:

* Person subject to a legal protection measure
* Vulnerable population: minors, persons under guardianship or trusteeship or persons deprived of their rights to liberty by court order.
* women with a known pregnancy
* Inability or refusal to comply with research requirements
* Active or weaned smoker > 15 PA
* Treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or opioids in the 10 days prior to inclusion

Case patient with asthma:

- Coexistence of a chronic inflammatory disease other than asthma

Case healthy volunteers:

- Coexistence of an inflammatory pathology

Exclusion criteria:

Cases asthma: Pregnancy during follow-up Cases healthy volunteers: Total IgE level greater than 100 kU/L (measured on the study sample)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Changes in expression of one or more molecules on the surface of NK cells | day 1 to day 2555
  Rationale for choice of primary endpoint: Our aim is to phenotype NK cells in different groups of severe asthma patients compared with control subjects, in order to identify at least one marker of disease discrimination on these cells. We are therefore looking for previously unknown changes in the expression of one or more molecules.

SECONDARY OUTCOMES:
Measurement of NK cell activation | day 1 to day 2555
  Change From Baseline in the expression of CD107, CD69 and interferon-ɣ.
Measurement of NK cell-induced epithelial cell activation and viability | day 1 to day 2555
  Change From Baseline in epithelial cell cohesion, mucin and cytokine (IL-8, type I interferon, IL-33 and TSLP) production

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital NORD - AP-HM, Clinique des bronches, de l'allergie et du sommeil, Marseille, France

IPD SHARING:
Plan to Share IPD: No